CLINICAL TRIAL: NCT00760032
Title: Association of Serum Levels of Lipopolysaccharide Binding Protein (LBP) With the Evolution of Pro- and Anti-inflammatory Cytokines, and the Development of Severe Infectious Events in Cirrhotic Patients
Brief Title: Lipopolysaccharide Binding Protein and Development of Infectious Events in Cirrhotic Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: was not possible to measure LBP levels because we cannot found the kit
Sponsor: Florencia Vargas-Vorackova (Other)
Collaborators: Laboratorios Senosiain, S.A. de C.V. (Industry)
Responsible Party: Sponsor-Investigator, Florencia Vargas-Vorackova, Doctor, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Organization: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: GAS-149-07-09-1; REF. 1612
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2012-12-05 (Estimated); Status verified 2012-12

CONDITIONS: Cirrhosis; Ascites; Infections
Keywords: Cirrhosis; Ascites; Lipopolysaccharide binding protein; Infections; Cytokines; Ciprofloxacin
MeSH Terms: conditions — Fibrosis; Ascites; Infections | interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): Ciprofloxacin
  Interventions: Drug: Ciprofloxacin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciprofloxacin — Ciprofloxacin oral, 500 mg capsules, one capsule per day during four weeks.
  Other Names: Ciproflox
  Arms: Active
Drug: Placebo — Placebo capsules, one capsule per day during four weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether plasma levels of lipopolysaccharide binding protein (LBP) are correlated with PBMN pro- and anti-inflammatory cytokine secretion, as well as with the development of severe infectious events in cirrhotic patients with ascites. As a secondary purpose, the study will evaluate the effect of a prophylactic administration of ciprofloxacin on LBP, cytokines and infections in the same patients.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis
* Ascites
* No history of spontaneous bacterial peritonitis and/or < 1 g of protein in ascites
* No antibiotic use in previous 6 weeks
* Absence of infection (documented by clinical history, blood cytology, urinalysis and urine culture, thorax x-ray and paracentesis)
* Absence of GI bleeding or encephalopathy
* Signature of informed consent

Exclusion Criteria:

* Ciprofloxacin contraindication
* Autoimmune hepatitis, sclerosing cholangitis or other autoimmune disease
* > 13 Child-Pugh points
* Inability to attend to regular visits
* Current alcohol intake
* Terminal disease with < 24 week expected survival

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Lipopolysaccharide binding protein plasma levels | 24 weeks

SECONDARY OUTCOMES:
Severe infection | 24 weeks
Pro- and anti-inflammatory cytokine secretion by PBMN cells | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Florencia Vargas-Vorackova, M.D., Ph.D., Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, México, D.f., Mexico

REFERENCES:
- See also: Sponsor's Web site — http://www.innsz.mx